CLINICAL TRIAL: NCT06544798
Title: Long-term Follow-up of AAV2-hAQP1 Gene Therapy in Participants With Radiation-Induced Late Xerostomia
Brief Title: Long-term Follow-up of Gene Therapy for Radiation-Induced Xerostomia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: MeiraGTx, LLC (Industry)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGT-AQP1-202
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Grade 2 and 3 Late Xerostomia Caused by Radiotherapy for Cancers of the Upper Aerodigestive Tract, Excluding the Parotid Glands
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the follow-up group or active treatment group based on the group to which they were randomized in Study MGT-AQP1-201.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Follow-up group (No Intervention): Participants who were randomized to AAV2-hAQP1 treatment in Study MGT-AQP1-201 will continue in this long-term follow-up schedule to complete an additional 48 months of follow-up after their end-of-study visit in Study MGT-AQP1-201. All study participants are to be followed for a period of 60 months after vector administration.
- Active treatment group (Experimental): Participants who were randomized to placebo treatment in Study MGT-AQP1-201, will be offered to transition from the long-term follow-up schedule to an active treatment schedule at the time of unblinding. Study drug administration should be completed after unblinding and after confirmation of the participant's continued eligibility for treatment. Upon completion of the 12-month primary treatment period, participants will continue in the study according to a follow-up schedule, to complete a total of 60 months of follow-up after AAV2-hAQP1 administration.
  Interventions: Genetic: AAV2-hAQP1

INTERVENTIONS:
Genetic: AAV2-hAQP1 — Administration of a prespecified concentration of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Arms: Active treatment group

SUMMARY:
This study will assess the long-term safety and efficacy of bilateral intra-parotid administration of AAV2-hAQP1 in adults with Grade 2 or Grade 3 radiation-induced late xerostomia.

DETAILED DESCRIPTION:
Individual participation in this study will last approximately 48 months for participants who received AAV2-hAQP1 in Study MGT-AQP1-201 and at least 60 months for participants who receive AAV2-hAQP1 in Study MGT-AQP1-202.

ELIGIBILITY:
Inclusion Criteria:

* Received study drug in Study MGT-AQP1-201

Exclusion Criteria:

* Withdrew consent to participate in Study MGT-AQP1-201.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with study drug-related adverse events and serious adverse events | From study start until Month 60 post-treatment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Miami Cancer Institute at Baptist Health South Florida, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Missouri, Columbia, Missouri
  - Erie County Medical Center, Buffalo, New York
  - Atrium Health, Charlotte, North Carolina
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
- Shirley and Jim Fielding Northeast Cancer Centre - Health Sciences North, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No